CLINICAL TRIAL: NCT04263623
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess the Efficacy and Safety of AT-5214 in the Treatment of Subjects With Moderate to Severe Palmar Hyperhidrosis
Brief Title: Clinical Study to Assess the Efficacy and Safety of AT-5214 in the Treatment of Subjects With Palmar Hyperhidrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atacama Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-9951-202
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Hyperhidrosis; Palmar Hyperhidrosis
Keywords: sweaty palms
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose (4 mg) (Experimental): Oral tablet containing 2 mg of active drug, dexmecamylamine HCl. Subjects will be instructed to take two tablets by mouth twice daily (in the morning and evening).
  Interventions: Drug: Dexmecamylamine HCl
- Low Dose (2 mg) (Experimental): Oral tablet containing 1 mg of active drug, dexmecamylamine HCl. Subjects will be instructed to take two tablets by mouth twice daily (in the morning and evening).
  Interventions: Drug: Dexmecamylamine HCl
- Placebo (Placebo Comparator): Oral tablet containing no active drug. Subjects will be instructed to take two tablets by mouth twice daily (in the morning and evening).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmecamylamine HCl — Investigational drug
  Other Names: AT-5214
  Arms: High Dose (4 mg); Low Dose (2 mg)
Other: Placebo — Oral tablet containing no active drug.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group comparison study of AT-5214 in subjects with moderate to severe primary palmar hyperhidrosis (sweaty palms). This study will compare two different oral (tablet) doses of AT-5214 (study drug) versus a matched placebo. Approximately 120 subjects will be enrolled at approximately 10 study sites.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of primary hyperhidrosis of the palms
* Subject is currently drug-naïve for hyperhidrosis medications
* Females must be post-menopausal, surgically sterile, or use an effective method of birth control

Exclusion Criteria:

* Subject is pregnant, lactating, is planning to become pregnant during the study, or is less than one year postpartum.
* Subject is a user of nicotine products within one year prior to Visit 1/Screening.
* Subject has known history of secondary hyperhidrosis.
* Subject has existence of neurological, psychiatric, endocrine, or other disease that can cause secondary hyperhidrosis or affect sweating.
* Subject has known history of Sjögren's syndrome or Sicca syndrome.
* Subject has used any of the following hyperhidrosis medications or therapies within the specified timeframe:

  1. Iontophoresis to the palms within four weeks prior to baseline visit;
  2. Botulinum toxin to the palms within one year prior to baseline visit;
  3. Prior surgical procedures to the palms (e.g., sympathectomy, debulking of sweat glands);
  4. Prior medical device treatment to the palms (approved or investigational);
  5. Any prescription treatments for hyperhidrosis within four weeks prior to baseline visit.
  6. Any topical antiperspirant treatment to the palms within 7 days prior to baseline visit.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has previously participated in a clinical study of dexmecamylamine or TC-5214.
* Subject has used an investigational drug or investigational device treatment within 30 days prior to baseline.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
PHIS Reduction | Week 6 (End of Study)
  Proportion of subjects with at least a 2-point reduction in the Palmar Hyperhidrosis Impact Scale (PHIS) from their mean baseline value (rated on an 11-point scale, 0-10).

SECONDARY OUTCOMES:
Absolute change in PHIS | Week 6 (End of Study)
  Absolute change from the mean baseline value in PHIS
Change in Sweat Production | Week 6 (End of Study)
  Proportion of subjects with a ≥50% reduction from the mean baseline value in gravimetrically measured sweat production.
Absolute change of Sweat Production | Week 6 (End of Study)
  Absolute change from mean baseline value in gravimetrically measured sweat production.

OTHER OUTCOMES:
Number of Subjects with Adverse Events (AEs) | Baseline (Day 1) to End of Study (Day 43)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No